CLINICAL TRIAL: NCT02906254
Title: Early Discontinuation of Empirical Antibacterial Therapy in Febrile Neutropenia: Prospective Observational Study (ANTIBIOSTOP)
Brief Title: Early Antibiotic Discontinuation in FUO
Acronym: ANTIBIOSTOP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ANTIBIOSTOP
Record Dates: First submitted 2016-09-02; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Febrile Neutropenia; Hematological Malignancy
MeSH Terms: conditions — Febrile Neutropenia; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ECIL-4 guidelines group: For the FUO group, antibiotics were stopped based on two procedures, irrespective of the neutrophil count or expected duration of neutropenia:
  - From 1st February 2014 to 30th November 2014, antibiotics were stopped when patients had been afebrile for more than 48 hours, as recommended by the ECIL-4 guidelines
  Interventions: Other: ECIL-4 guidelines group
- short-course antibiotic therapy: For the FUO group, antibiotics were stopped based on two procedures, irrespective of the neutrophil count or expected duration of neutropenia:
  - From 1st December 2014 to 30th September 2015, antibiotics were stopped on day 5 in febrile or afebrile patients (short-course antibiotic therapy).
  Interventions: Other: ECIL-4 guidelines group; Other: Short-course antibiotic therapy

INTERVENTIONS:
Other: ECIL-4 guidelines group — Antibiotics were stopped when patients had been afebrile for more than 48 hours
Other: Short-course antibiotic therapy — Antibiotics were stopped on day 5 in febrile or afebrile patients
  Groups: short-course antibiotic therapy

SUMMARY:
Febrile neutropenia requires prompt initiation of broad-spectrum antibiotics, which can be responsible for side-effects and selection of resistance. This study demonstrates the safety of an early discontinuation of empirical treatments, in carefully selected patients presenting with fever of unknown origin.

DETAILED DESCRIPTION:
Infections are responsible for significant morbidity and mortality in haematological patients, in particular during chemotherapy-induced neutropenia. Guidelines recommend immediate initiation of antibiotic therapy, whose optimal duration is unclear. The primary objective of this study is to evaluate early discontinuation of antibiotic treatment for Fever of Unknown Origin (FUO) in afebrile or febrile neutropenic patients. The secondary objective is to describe the epidemiology of febrile neutropenia (FN) in investigator centre.

Every episode of FN was prospectively identified. In the first phase of the study, empirical antibiotic therapy of FUO patients was stopped after 48 hours of apyrexia, in accordance with ECIL-4 (European Conference on Infections in Leukaemia) recommendations. In the second phase of the study, antibiotics were stopped on day 5 for all FUO patients, regardless of their temperature or their leukocyte count.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* presence of a malignant haematological disease combined with chemotherapy-induced neutropenia (polymorphonuclear neutrophil (PMN) count ≤ 500/mm3)
* fever defined by tympanic temperature of ≥38°C for ≥1 hour or a single temperature of ≥38.3°C

Exclusion Criteria:

* Patients without curative care
* chronic neutropenia (PMN≤ 500/mm3 for 3 months or more)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient admitted to the Department of Clinical Haematology of Brest Teaching Hospital (France) was eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety of a short-term antibiotic treatment in afebrile or febrile patients exhibiting FUO, irrespective of their neutrophil count. | Month 1
  mortality, intensive care admissions, infection
tolerability of a short-term antibiotic treatment in afebrile or febrile | Month 1
  Duration of antibiotic therapy (days), duration of fever (days)

SECONDARY OUTCOMES:
Epidemiology of febrile neutropenia | Month 1
  Clinical and biological data

CONTACTS AND LOCATIONS:
Overall Officials: Gaelle Guillerm, MD, Principal Investigator — Department of Hematology, Brest Teaching Hospital, Hospital Morvan, Avenue Foch, 29200 Brest, France; Jean-Philippe Talarmin, MD, Principal Investigator — Department of Internal Medicine, Infectious Diseases and Hematology, Cornouaille Hospital Quimper, Avenue Yves Thépot, 29000 Quimper, France; Lenaïg Le Clech, MD, Principal Investigator — Department of Hematology, Brest Teaching Hospital, Hospital Morvan, Avenue Foch, 29200 Brest, France
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided